CLINICAL TRIAL: NCT00535886
Title: The Effects of Natural Versus Man-Made Trans Fatty Acids on Lipoprotein Profiles: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MM6222; IRB# 2005-45
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2007-09

CONDITIONS: Cardiovascular Disease; Diabetes; Dyslipidemia
Keywords: Trans Fatty Acids; conjugated linoleic acid; vaccenic acid; High Density Lipoprotein Cholesterol; Low Density Lipoprotein Cholesterol; Beef
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Dyslipidemias | interventions — Oleic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Elaidic Acid (Active Comparator)
  Interventions: Dietary Supplement: Man-made Trans FA
- Vaccenic Acid (Experimental)
  Interventions: Dietary Supplement: Natural Trans FA
- Oleic Acid (Placebo Comparator)
  Interventions: Dietary Supplement: Oleic Acid

INTERVENTIONS:
Dietary Supplement: Man-made Trans FA — EA as 6% of total energy
  Arms: Elaidic Acid
Dietary Supplement: Natural Trans FA — VA as 6% of total energy
  Arms: Vaccenic Acid
Dietary Supplement: Oleic Acid — OA as 6% of total energy
  Arms: Oleic Acid

SUMMARY:
The purpose of this study is to test the effects of natural vs. man-made trans fatty acids (trans fats) on blood cholesterol.

DETAILED DESCRIPTION:
Since the purpose of the study is to determine the statistical power required for a definitive study testing and comparing the effects of two trans fatty acids, vaccenic and elaidic acid, on lipoprotein profiles, no hypotheses will be specified.

Specific Aims:

1. To determine the variability in the lipid and lipoprotein response to diets enriched in natural versus man-made trans fats in order to appropriately power a larger scale clinical study
2. To optimize the delivery of trans fat-enriched diets through the development of supplemental food items

The adverse health effects of trans fatty acids (TFA) on cardiovascular disease (CVD) risk have been established in a number of metabolic and epidemiological studies [Willett 1993, Hu 1997, Ascherio 1996, Pietinen 1997, Oomen 2001]. Trans fats are fatty acids with 18 carbon chains and one or more double bond(s). The hydrogen atoms of the double bond(s) are in a configuration (trans rather than cis) that results in the straightening of a normally kinked unsaturated fatty acid chain. Trans fats occur naturally in low quantities in dairy and beef products, but have also been artificially introduced to the food supply by the process of the hydrogenation of vegetable oils [Mann 1994]. Only two studies linking the consumption of trans fatty acids with an increased risk of CVD have distinguished between the effects of man-made versus naturally occurring trans fatty acids [Willett 1993, Oomen 2001].

It has been suggested that the relationship between trans fatty acids and coronary heart disease is specifically attributable to man-made trans fatty acids. In fact, some of the trans fats that occur naturally in animal products, in particular, conjugated linoleic acid (CLA), may have beneficial health effects. CLA has been shown to be anti-carcinogenic [Ip 2003], anti-atherogenic [McLeod 2004] and anti-diabetic [Rainer 2004]; it has also been shown to enhance the immune response and have positive effects on growth and energy partitioning. As a precursor to CLA, vaccenic acid (VA), another trans fatty acid found in dairy and beef products, may also provide health benefits. Bioconversion of VA to CLA has been recently demonstrated [Turpeinen 2002]. The effects of diet supplementation with VA on health parameters have yet to be defined.

The objective of the overall research project will be to test the hypothesis that the ingestion of high doses of naturally occurring VA does not cause the adverse lipid and lipoprotein effects known to occur with the consumption of man made trans fatty acids, in particular, elaidic acid (EA). The latter is the primary trans fatty acid found in products such as margarines, cakes, cookies, crackers and other baked and processed foods [Steinhart 2003]. The primary outcome measure will be the ratio of total to high density lipoprotein (HDL) cholesterol. Related secondary outcome measures include concentrations of low density lipoprotein (LDL) cholesterol, HDL cholesterol, triglyceride (TG) and Lp(a). The present proposal is designed to test the feasibility of, and determine the power for, a definitive study.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age >= 18 years
* Body mass index (BMI) less than 35 kg/m*m
* Fasting total cholesterol and LDL cholesterol less than the 95% for age and sex
* Fasting triglyceride <= 400 mg/dl
* Fasting blood glucose <= 125 mg/dl
* Fasting thyroid stimulating hormone less than 0.3 or greater than 5.0 uIU/ml
* Blood pressure <= 150/90
* Agrees to no alcohol during the study
* Agrees to maintain same level of physical activity throughout the study

Exclusion Criteria:

* Smokers
* Personal history of coronary heart disease, cerebrovascular disease or vascular disease, diabetes, bleeding disorder, liver or renal disease, or of cancer (other than skin cancer) in the last five years.
* Use of drugs known to affect lipid metabolism, blood thinning agents, or hormones.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-11; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the ratio of total to high density lipoprotein (HDL) cholesterol. Blood draws will take place at screening, three weeks, and five weeks. | Five weeks

SECONDARY OUTCOMES:
Related secondary outcome measures include concentrations of low density lipoprotein (LDL) cholesterol, HDL cholesterol, triglyceride (TG) and Lp(a) measured at screening, three weeks, and five weeks. | Five weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, M.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland; Patty Siri, Ph.D., Study Director — UCSF Benioff Children's Hospital Oakland; Shira Miller, M.D., Study Director — National Cattlemen's Beef Association, a contractor to the Beef Checkoff
Locations (1):
- Children's Hospital Oakland Research Institute, Oakland, California, United States

REFERENCES:
- [Background] Willett WC, Stampfer MJ, Manson JE, Colditz GA, Speizer FE, Rosner BA, Sampson LA, Hennekens CH. Intake of trans fatty acids and risk of coronary heart disease among women. Lancet. 1993 Mar 6;341(8845):581-5. doi: 10.1016/0140-6736(93)90350-p. PMID 8094827
- [Background] Hu FB, Stampfer MJ, Manson JE, Rimm E, Colditz GA, Rosner BA, Hennekens CH, Willett WC. Dietary fat intake and the risk of coronary heart disease in women. N Engl J Med. 1997 Nov 20;337(21):1491-9. doi: 10.1056/NEJM199711203372102. PMID 9366580
- [Background] Ascherio A, Rimm EB, Giovannucci EL, Spiegelman D, Stampfer M, Willett WC. Dietary fat and risk of coronary heart disease in men: cohort follow up study in the United States. BMJ. 1996 Jul 13;313(7049):84-90. doi: 10.1136/bmj.313.7049.84. PMID 8688759
- [Background] Pietinen P, Ascherio A, Korhonen P, Hartman AM, Willett WC, Albanes D, Virtamo J. Intake of fatty acids and risk of coronary heart disease in a cohort of Finnish men. The Alpha-Tocopherol, Beta-Carotene Cancer Prevention Study. Am J Epidemiol. 1997 May 15;145(10):876-87. doi: 10.1093/oxfordjournals.aje.a009047. PMID 9149659
- [Background] Oomen CM, Ocke MC, Feskens EJ, van Erp-Baart MA, Kok FJ, Kromhout D. Association between trans fatty acid intake and 10-year risk of coronary heart disease in the Zutphen Elderly Study: a prospective population-based study. Lancet. 2001 Mar 10;357(9258):746-51. doi: 10.1016/s0140-6736(00)04166-0. PMID 11253967
- [Background] Mann GV. Metabolic consequences of dietary trans fatty acids. Lancet. 1994 May 21;343(8908):1268-71. doi: 10.1016/s0140-6736(94)92157-1. PMID 7910281
- [Background] Ip MM, Masso-Welch PA, Ip C. Prevention of mammary cancer with conjugated linoleic acid: role of the stroma and the epithelium. J Mammary Gland Biol Neoplasia. 2003 Jan;8(1):103-18. doi: 10.1023/a:1025739506536. PMID 14587866
- [Background] McLeod RS, LeBlanc AM, Langille MA, Mitchell PL, Currie DL. Conjugated linoleic acids, atherosclerosis, and hepatic very-low-density lipoprotein metabolism. Am J Clin Nutr. 2004 Jun;79(6 Suppl):1169S-1174S. doi: 10.1093/ajcn/79.6.1169S. PMID 15159253
- [Background] Rainer L, Heiss CJ. Conjugated linoleic acid: health implications and effects on body composition. J Am Diet Assoc. 2004 Jun;104(6):963-8, quiz 1032. doi: 10.1016/j.jada.2004.03.016. PMID 15175596
- [Background] Turpeinen AM, Mutanen M, Aro A, Salminen I, Basu S, Palmquist DL, Griinari JM. Bioconversion of vaccenic acid to conjugated linoleic acid in humans. Am J Clin Nutr. 2002 Sep;76(3):504-10. doi: 10.1093/ajcn/76.3.504. PMID 12197992
- [Background] Steinhart H, Rickert R, Winkler K. Trans fatty acids (TFA): analysis, occurrence, intake and clinical relevance. Eur J Med Res. 2003 Aug 20;8(8):358-62. PMID 12915330
- [Background] Griinari JM, Corl BA, Lacy SH, Chouinard PY, Nurmela KV, Bauman DE. Conjugated linoleic acid is synthesized endogenously in lactating dairy cows by Delta(9)-desaturase. J Nutr. 2000 Sep;130(9):2285-91. doi: 10.1093/jn/130.9.2285. PMID 10958825